CLINICAL TRIAL: NCT07023978
Title: Effects of Qigong on General Well-being, Anxiety, and Physical Activity in Pregnant Women
Brief Title: on General Well-being, Anxiety, and Physical Activity in Pregnant Women
Acronym: Qigong
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Emine Dundar Ahi, MD, Physical medicine and rehabilitation specialist, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA24/178; Emine Ahi (Other: Private clinic)
Record Dates: First submitted 2025-06-01; First posted 2025-06-17 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy
MeSH Terms: interventions — Movement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control arm (No Intervention): 50 Pregnant women in the control group will be given pregnancy counseling that includes only nutrition, walking (3 days a week for 30 minutes), and breathing exercises, and will be called for 1st, 2nd and 3rd month check-ups.
- Qigong arm (Active Comparator): In addition to pregnancy counseling, the Qigong group will receive (52 participants) 2 Qigong training sessions, one via Zoom and one face-to-face, and then the training videos of each exercise will be sent via WhatsApp. Patients will be asked to do the Qigong exercises at home for 30 minutes, 3 days a week for 12 weeks. These patients will be called for 1-month, 2-month and 3-month check-ups.
  Interventions: Other: Some movements in the qigong study called Ba Duan Jin, which will be applied to pregnant women, will be arranged for pregnant women and explained in detail. These are very slow, movements

INTERVENTIONS:
Other: Some movements in the qigong study called Ba Duan Jin, which will be applied to pregnant women, will be arranged for pregnant women and explained in detail. These are very slow, movements — Ba Duan Jin Qigong
  Arms: Qigong arm

SUMMARY:
102 pregnant women will be randomly divided into 2 groups. Participants in the control group will be given pregnancy counseling that includes only nutrition, walking (3 days a week for 30 minutes), and breathing exercises, and will be called for 1st, 2nd and 3rd month check-ups. In addition to pregnancy counseling, the Qigong group will receive 2 Qigong training sessions, one via Zoom and one face-to-face, and then the training videos of each exercise will be sent via WhatsApp. Paricipants will be asked to do the Qigong exercises at home for 30 minutes, 3 days a week for 12 weeks. These participants will be called for 1-month, 2-month and 3-month check-ups. Blood pressure and sugar measurements will be recorded at the first visit, 1st month, 2nd month and 3rd month check-ups, and patients will also be evaluated with the Pregnancy Physical Activity Questionnaire, Pregnancy Stress Assessment Scale, Pregnancy-related Anxiety Scale, Pregnancy Exercise Self-Efficacy Questionnaire. After the recruitment period the results will be evaluated statistically.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-40 who have a new pregnancy detected by USG
* Pregnant women whose pregnancy week is compatible with fetal development, who do not have any problems and who will not have any problems exercising

Exclusion Criteria:

* Those with risky pregnancies (cervical dilation, bleeding, premature membrane rupture, etc.) *<18 and >40 years old pregnant women

  * Those with cardiovascular disease or hypertension
  * Those with uncontrolled diabetes
  * Those with uncontrolled thyroid disease
  * Those with a previous risky pregnancy or a complication
  * Those with an operation, metabolic bone disease or joint limitation that will prevent them from exercising
  * Those who are included in another pregnancy counseling or physical activity program
  * Those who do not give their consent for the study, do not come to regular pregnancy check-ups or have incomplete information will be excluded from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy females will be participate
Enrollment: 102 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Values | 2 minutes
  Glucose is the key metabolic substrate for tissue energy production. In the perinatal period the mother supplies glucose to the fetus and for most of the gestational period the normal lower limit of fetal glucose concentration is around 3 mmol/L. diabetes is high blood sugar (glucose) that develops during pregnancy and usually disappears after giving birth. It can happen at any stage of pregnancy, but is more common in the second or third trimester.
Pregnancy Exercise Self-Efficacy Scale | 10 minutes
  The Pregnancy Exercise Self-Efficacy Scale (P-ESES) is a validated tool designed to assess a pregnant woman's confidence in her ability to engage in physical activity during pregnancy. It measures self-efficacy across various situations that may influence exercise behavior, such as fatigue, lack of time, or discomfort. The scale typically includes a set of statements where respondents rate their confidence levels using a Likert-type scale (usually from 1 = not at all confident to 5 = completely confident). Higher total scores indicate greater self-efficacy regarding exercise during pregnancy. The final score is calculated by summing all item responses, and it helps identify women who may need additional support or encouragement to stay active.
blood pressure value | 2 minutes
  High blood pressure during pregnancy occurs when a pregnant woman has a blood pressure reading of 140/90 mm Hg or higher in two readings that are 4 or more hours apart. Severe high blood pressure during pregnancy occurs when a pregnant woman has a blood pressure reading of 160/110 mm Hg on two or more occasions

SECONDARY OUTCOMES:
The 30-item Pregnancy Stress Rating Scale (PSRS) | 10 minutes
  The PSRS36 is a psychometrically sound and practical tool for nurses and other healthcare providers to assess prenatal stress and to examine intervention protocols in Taiwanese prenatal women. More research is recommended to determine whether the PSRS36 may be used in other racial-ethnic groups.
Pregnancy-related anxiety scale | 10 minutes
  Pregnancy-related anxiety is a specific anxiety characterized by fears and worries about pregnancy. This distinct anxiety is associated with various adverse neonatal (e.g., preterm birth), obstetric (e.g., prolonged and difficult labor), and maternal outcomes (e.g., mood disorders). While several scales exist that assess pregnancy-related anxiety, there is limited information on their development and psychometric properties. Moreover, general anxiety scales used to assess anxiety in pregnant women can confound assessment by the similarity of common pregnancy experiences with anxiety symptomology (e.g., poor sleep). The development of the Pregnancy-related Anxiety Scale (PrAS) addressed this gap, and since its development, the PrAS has demonstrated sound psychometric properties. To meet antenatal anxiety-screening guidelines that advocate using brief scales, the PrAS was refined to a 15-item version. To

CONTACTS AND LOCATIONS:
Locations (1):
- Home adress of the principal investigator, Kocaeli, Turkey (Türkiye)